CLINICAL TRIAL: NCT04850417
Title: Randomized Clinical Trial Assessing the Value of Beta-Blockers and Antiplatelet Agents in Patients With Spontaneous Coronary Artery Dissection. (The BA-SCAD Randomized Clinical Trial)
Brief Title: Randomized Study of Beta-Blockers and Antiplatelets in Patients With Spontaneous Coronary Artery Dissection
Acronym: BA-SCAD
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Spanish Society of Cardiology (Other)
Collaborators: Instituto de Investigación Sanitaria Hospital Universitario de la Princesa (Other); Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Responsible Party: Principal Investigator, Fernando Alfonso, Principal Investigator, Spanish Society of Cardiology
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: BA-SCAD
Record Dates: First submitted 2021-04-07; First posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Spontaneous Coronary Artery Dissection
Keywords: Spontaneous coronary artery dissection; Beta-blockers; Antiplatelets; Coronary angiography; Intracoronary imaging; Biomarkers; Myocardial infarction
MeSH Terms: conditions — Coronary Artery Dissection, Spontaneous; Myocardial Infarction | interventions — Adrenergic beta-Antagonists; Aspirin; Clopidogrel

STUDY DESIGN:
Intervention Model Description: Factorial 2x2 design (a) beta-blockers yes/no; b) Antiplatelets short/long)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Beta-blockers and Short Antiplatelet Therapy (Experimental): Beta-blockers (experimental) and Short Antiplatelet Therapy (experimental). Aspirin alone recommended for Short Antiplatelet Therapy
  (The main comparison of this randomized clinical trial (2x2, factorial design) is beta-blockers vs no beta-blockers and short vs long-term antiplatelet therapy)
  Interventions: Drug: Beta blocker, aspirin, clopidogrel
- Beta-blockers and Long Antiplatelet Therapy (Experimental): Beta-blockers (experimental) and Long Antiplatelet Therapy. Aspirin and Clopidogrel recommended in Long Antiplatelet Therapy
  (The main comparison of this randomized clinical trial (2x2, factorial design) is beta-blockers vs no beta-blockers and short vs long-term antiplatelet therapy)
  Interventions: Drug: Beta blocker, aspirin, clopidogrel
- No Beta-blockers and Short Antiplatelet Therapy (Experimental): No Beta-blockers and Short Antiplatelet Therapy (experimental). Aspirin alone recommended in Short Antiplatelet Therapy
  (The main comparison of this randomized clinical trial (2x2, factorial design) is beta-blockers vs no beta-blockers and short vs long-term antiplatelet therapy)
  Interventions: Drug: Beta blocker, aspirin, clopidogrel
- No Beta-blockers and Long Antiplatelet Therapy (Active Comparator): No Beta-blockers and Long Antiplatelet Therapy. Aspirin and Clopidogrel recommended in Long Antiplatelet Therapy
  (The main comparison of this randomized clinical trial (2x2, factorial design) is beta-blockers vs no beta-blockers and short vs long-term antiplatelet therapy)
  Interventions: Drug: Beta blocker, aspirin, clopidogrel

INTERVENTIONS:
Drug: Beta blocker, aspirin, clopidogrel — Pragmatic design. Beta-blockers and Antiplatelets drugs selected by the investigators. Asprin and Clopidogrel recomended for patients allocated to prologed DAPT. Aspirin Alone recomended for patients allocated to short antiplatelet therapy
  Other Names: Beta-blockers; Aspirin; Clopidogrel

SUMMARY:
Spontaneous coronary artery dissection (SCAD) is a cause of acute coronary syndrome (ACS). Most patients are treated with beta-blockers (BB) and antiplatelet drugs (AP) on empiric basis. The Beta-Blockers and Antiplatelet Agents in Patients with Spontaneous Coronary Artery Dissection (BA-SCAD) randomized clinical trial is an academic, pragmatic, nation-wide, prospective study developed under the auspices of the Spanish Society of Cardiology (SEC) that aims to assess the efficacy of medical therapy in SCAD patients. Using a factorial 2x2 design, patients will be randomized (1:1/1:1) to: 1) BB (yes/no) and 2) short AP regimen (1 month) vs prolonged dual AP therapy (DAPT) (12 months).Only patients with preserved left ventricular ejection fraction (LVEF) will be randomized to BB (yes/no) because patients with LVEF <40% will receive BB according to current guidelines. Likewise, only medically managed patients will be randomized to short AP therapy vs 1-year DAPT. The study will have a pragmatic, open label, blind outcomes design (PROBE). A total of 600 SCAD patients will be randomized within 2 years (300 per arm in a factorial 2x2 design). The primary efficacy endpoint will include the composite of death, acute myocardial infarction (MI), stroke, coronary revascularization, recurrent SCAD, and unplanned hospitalization for ACS or heart failure at 1 year. The primary safety endpoint will be bleeding. All patients will be clinically followed yearly. The main study will be pragmatic but a comprehensive set of additional studies (clinical, imaging, biomarkers, inflammatory, immunologic, pharmacogenetic and genetic) will be organized to ensure an holistic view on this challenging condition.

DETAILED DESCRIPTION:
Spontaneous coronary artery dissection (SCAD) is a relatively rare but important and increasingly recognized cause of acute coronary syndrome (ACS). Most patients presenting with SCAD are treated with beta-blockers (BB) and antiplatelet drugs (AP). Although appealing from a pathophysiological standpoint, such management strategy is completely empiric. The Beta-Blockers and Antiplatelet Agents in Patients with Spontaneous Coronary Artery Dissection (BA-SCAD) randomized clinical trial is an academic, pragmatic, nation-wide, prospective study developed under the auspices of the Spanish Society of Cardiology (SEC) that aims to assess the efficacy of medical therapy in SCAD patients. Using a factorial 2x2 design, patients will be randomized (1:1/1:1) to: 1) BB (yes/no) and 2) short AP regimen (1 month) vs prolonged dual AP therapy (DAPT) (12 months). A conservative medical management will be initially recommended, with coronary revascularization reserved for patients with ongoing/refractory ischemia. Only patients with preserved left ventricular ejection fraction (LVEF) will be randomized to BB (yes/no) because patients with LVEF <40% will receive BB according to current guidelines. Likewise, only medically managed patients will be randomized to short AP therapy vs 1-year DAPT, because patients requiring coronary interventions will receive DAPT. The study will have a pragmatic, open label, blind outcomes design (PROBE). The type and dose of BB and AP agents will be at the discretion of the treating physician. Treatment adherence will be reinforced and closely monitored and the potential influence of drug discontinuation/cross-over on outcomes will be carefully evaluated. A total of 600 SCAD patients will be randomized within 2 years (300 per arm in a factorial 2x2 design). The primary efficacy endpoint will include the composite of death, acute myocardial infarction (MI), stroke, coronary revascularization, recurrent SCAD, and unplanned hospital admission for ACS or heart failure at 1 year. The primary safety endpoint will be bleeding according the Bleeding Academic Research Consortium (BARC) criteria ≥ 3. An analysis of net clinical benefit, including primary efficacy and safety endpoints, will also be performed. All patients will be clinically followed at 1 year (primary endpoint) and yearly thereafter. Although the main study will be pragmatic, following routine clinical practice, a systematic and comprehensive set of additional ancillary studies and investigations (clinical, imaging, biomarkers, inflammatory, immunologic, pharmacogenetic and genetic) will be prospectively organized to ensure a multidisciplinary and holistic view on this challenging condition.

ELIGIBILITY:
Inclusion Criteria:

* Angiographic diagnosis of SCAD
* Admission for ACS or other manifestations of ischemia
* Informed consent

Exclusion Criteria:

* Cardiogenic shock or severe hemoynamic instability
* Concomitant severe heart disease requiring surgical correction (in <2 years)
* Medical condition seriously limiting life expectancy (< 2 years)
* Allergies or contraindication to drugs required in one of the study arms; the patient may be randomized in the other arm (factorial design)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-04-30 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
MACE (death, myocardial infarction, coronary revascularization, recurrent SCAD, stroke, unplanned admission for heart failure or acute coronary syndrome with dynamic ECG changes) | 1 year
  MACE (death, myocardial infarction, coronary revascularization, recurrent SCAD, stroke, unplanned admission for heart failure or acute coronary syndrome with dynamic ECG changes)

SECONDARY OUTCOMES:
MACE (death, myocardial infarction, coronary revascularization, stroke and heart failure) | 1, 2 and 3 years
  MACE (death, myocardial infarction, coronary revascularization, stroke and heart failure)
MACE (death, myocardial infarction, coronary revascularization) | 1, 2 and 3 years
  MACE (death, myocardial infarction, coronary revascularization)
MACE (death, myocardial infarction) | 1, 2 and 3 years
  MACE (death, myocardial infarction)
MACE (death, myocardial infarction, coronary revascularization, recurrent SCAD, stroke, unplanned admission for heart failure or acute coronary syndrome with dynamic ECG changes) | 2, 3,4 and 5 years
  MACE (death, myocardial infarction, coronary revascularization, recurrent SCAD, stroke, unplanned admission for heart failure or acute coronary syndrome with dynamic ECG changes)
Safety: Major Bleeding | 1 year
  Major Bleeding (BARC >=3)
Safety: Bleeding | 1 year
  Bleeding (BARC >=2)
MACE and Bleeding | 1, 2 and 3 years
  MACE (death, myocardial infarction, coronary revascularization, recurrent SCAD, stroke, unplanned admission for heart failure or acute coronary syndrome with dynamic ECG changes) and bleeding
Death | 1, 2 and 3 years
  Death
Myocardial infarction | 1, 2 and 3 years
  Myocardial infarction
Coronary revascularization | 1, 2 and 3 years
  Coronary revascularization
Recurrent SCAD | 1, 2 and 3 years
  Recurrent SCAD
Stroke | 1, 2 and 3 years
  Stroke
Unplanned admission for heart failure | 1, 2 and 3 years
  Unplanned admission for heart failure
Unplanned admission for acute coronary syndrome with dynamic ECG changes | 1, 2, 3 years
  Unplanned admission for acute coronary syndrome with dynamic ECG changes

OTHER OUTCOMES:
Substudy on strategies and results of coronary interventions | Through study completion, up to 5 years
  Strategies and results of coronary interventions (different devices and modalities). Procedural success and angiographic results
Substudy on angiographic findings in relation to prognosis | Through study completion, up to 5 years
  Angiographic analysis (visual and QCA, central corelab). Quantitative coronary angiography analyses (MLD, % diameter stenosis, TIMI Flow)
Substudy on value of intracoronary imaging in SCAD (OCT and IVUS) | Through study completion, up to 5 years
  Intracoronary imaging in SCAD (central corelab) (OCT [optical coherence tomography] and IVUS [intravascular ultrasound] ). Minimal lumen area.
Non-invasive imaging techniques | Through study completion, up to 5 years
  Cardiac CT and CMR (coronary and peripheral arteries) (central corelab)
Substudy on inflammation and biomarkers | Through study completion, up to 5 years
  Comprehensive analysis of biomarkers. Coordinating center (HULP). Including leucocytes, HsCRP, IL6
Pharmacogenomic study | Through study completion, up to 5 years
  Pharmacogenomic study. Coordinating center (HULP). Percent of responders to treatment according to the pharmacogenomic profile
Micro RNAs and Genetic studies | Through study completion, up to 5 years
  Micro RNAs and Genetic studies. Coordinating center (HULP). Array of different micro-RNAs

CONTACTS AND LOCATIONS:
Overall Officials: Spanish Society of Cardiology Spanish Society of Cardiology, Study Chair — Spanish Society of Cardiology

IPD SHARING:
Plan to Share IPD: Yes
To be decided by the steering committee upon formal official request by academic investigators
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the primary endpoint is reported
Access Criteria: To be discussed

REFERENCES:
- [Derived] Alfonso F, de la Torre Hernandez JM, Ibanez B, Sabate M, Pan M, Gulati R, Saw J, Angiolillo DJ, Adlam D, Sanchez-Madrid F. Rationale and design of the BA-SCAD (Beta-blockers and Antiplatelet agents in patients with Spontaneous Coronary Artery Dissection) randomized clinical trial. Rev Esp Cardiol (Engl Ed). 2022 Jun;75(6):515-522. doi: 10.1016/j.rec.2021.08.003. Epub 2021 Sep 22. English, Spanish. PMID 34561195